CLINICAL TRIAL: NCT04303780
Title: A Phase 3 Multicenter, Randomized, Open Label, Active-controlled, Study of AMG 510 Versus Docetaxel for the Treatment of Previously Treated Locally Advanced and Unresectable or Metastatic NSCLC Subjects With Mutated KRAS p.G12C
Brief Title: Study to Compare AMG 510 "Proposed INN Sotorasib" With Docetaxel in Non Small Cell Lung Cancer (NSCLC) (CodeBreak 200).
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20190009; 2023-508214-42-00 (Other: CTIS (EU))
Expanded Access: NCT04667234 (No longer available)
Record Dates: First submitted 2020-03-05; First posted 2020-03-11 (Actual); Results first posted 2023-05-10 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: KRAS p, G12c Mutated /Advanced Metastatic NSCLC
MeSH Terms: interventions — sotorasib; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AMG 510 (Experimental)
  Interventions: Drug: AMG 510
- Docetaxel (Active Comparator)
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: AMG 510 — 21 day cycles
  Arms: AMG 510
Drug: Docetaxel — 21 day cycles
  Arms: Docetaxel

SUMMARY:
A Phase 3 Study to Compare AMG 510 with Docetaxel in Non Small Cell Lung Cancer (NSCLC) subjects with KRAS p. G12c mutation

ELIGIBILITY:
Inclusion Criteria:

* Men or women greater than or equal to 18 years old.
* ECOG ≤ 1
* Pathologically documented, previously treated, locally-advanced and unresectable or metastatic NSCLC with KRAS p.G12C mutation confirmed through central testing or have documentation of KRAS p.G12C mutation through Amgen Study 20190294 prior to enrollment

Exclusion Criteria:

* Active brain metastases
* Myocardial infarction within 6 months of study day 1
* Gastrointestinal (GI) tract disease causing the inability to take oral medication

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 345 (Actual)
Dates: Start 2020-06-04 (Actual); Primary Completion 2022-08-02 (Actual); Study Completion 2026-02-25 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (273):
- United States (53):
  - Pacific Cancer Medical Center Inc, Anaheim, California
  - City of Hope National Medical Center, Duarte, California
  - Pacific Shores Medical Group Long Beach, Long Beach, California
  - University of California Los Angeles, Los Angeles, California
  - University of California at Davis Medical Center, Sacramento, California
  - Ridley Tree Cancer Center, Santa Barbara, California
  - University of California San Francisco Mission Hall, Stanford, California
  - Harbor University of California Los Angeles Medical Center, Torrance, California
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Danbury Hospital, Norwalk, Connecticut
  - Medical Oncology Hematology Consultants Helen F Graham Cancer Center, Newark, Delaware
  - Washington Cancer Institute at MedStar Washington Hospital, Washington D.C., District of Columbia
  - Florida Cancer Specialists - Fort Myers, Fort Myers, Florida
  - Memorial Regional Hospital, Hollywood, Florida
  - Florida Cancer Specialists Research North, St. Petersburg, Florida
  - Florida Cancer Specialists Research Panhandle, Tallahassee, Florida
  - Emory University, Atlanta, Georgia
  - Northside Hospital, Incorporated, Atlanta, Georgia
  - Affiliated Oncologists, LLC, North Chicago, Illinois
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Willis Knighton Cancer Center, Shreveport, Louisiana
  - Maryland Oncology Hematology PA, Clinton, Maryland
  - New York Cancer and Blood Specialists, Lowell, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Center for Oncology Clinical Trials, Grand Rapids, Michigan
  - Minnesota Oncology Hematology PA, Minneapolis, Minnesota
  - HCA Midwest Health Kansas City, Kansas City, Missouri
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Summit Medical Group, Florham Park, New Jersey
  - New York Oncology Hematology, PC, Albany, New York
  - United States Oncology Regulatory Affairs Corporate Office, Albany, New York
  - Northwell Health Monter Cancer Center, Lake Success, New York
  - Montefiore Einstein Center for Cancer Care, The Bronx, New York
  - James J Peters VA Medical Center, The Bronx, New York
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Oncology Hematology Care Inc, Cincinnati, Ohio
  - Northwest Cancer Specialists - Vancouver, Portland, Oregon
  - Charleston Oncology, Charleston, South Carolina
  - Saint Francis Hospital, Inc, Greenville, South Carolina
  - Tennessee Oncology PLLC, Chattanooga, Tennessee
  - Tennessee Cancer Specialists, Knoxville, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - Texas Oncology-Bedford, Bedford, Texas
  - Texas Oncology Baylor, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - Valley Cancer Associates, Harlingen, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - US Oncology Research Investigational Products Center, Irving, Texas
  - Hope Cancer Center, Tyler, Texas
  - Intermountain Medical Center, Murray, Utah
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
- Australia (10):
  - Blacktown Hospital, Blacktown, New South Wales
  - Chris OBrien Lifehouse, Camperdown, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Prince Charles Hospital, Chermside, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - St John of God Healthcare, Subiaco, Western Australia
- Belgium (9):
  - Institute Jules Bordet, Brussels
  - Universite Catholique de Louvain Cliniques Universitaires Saint Luc, Brussels
  - Grand Hopital de Charleroi, Charleroi
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Universitair Ziekenhuis Gent, Ghent
  - Universitair Ziekenhuis Leuven - Campus Gasthuisberg, Leuven
  - Centre Hospitalier Universitaire de Liege, Liège
  - AZ Delta Campus Rumbeke, Roeselare
  - Algemeen Ziekenhuis Nikolaas Campus Sint Niklaas, Sint-Niklaas
- Brazil (10):
  - Hospital de Caridade de Ijui, Ijuí, Rio Grande do Sul
  - Hospital Sao Lucas da Pontificia Universidade Catolica do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Sociedade Beneficente de Senhoras Hospital Sirio Libanes, São Paulo, SÃ£o Paulo
  - Beneficencia Portuguesa de Sao Paulo, São Paulo, SÃ£o Paulo
  - Oncologia Rede DÂ´Or, São Paulo, SÃ£o Paulo
  - Hospital Israelita Albert Einstein, São Paulo, SÃ£o Paulo
  - Hospital de Base de Sao Jose do Rio Preto, SÃ£o JosÃ© Do Rio Preto, SÃ£o Paulo
  - Fundacao Antonio Prudente - Hospital A C Camargo, SÃ£o Paulo, SÃ£o Paulo
  - Centro de Tratamento de Tumores Botafogo, Rio de Janeiro
  - Instituto Coi, Rio de Janeiro
- Canada (7):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Juravinski Cancer Centre, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Centre Hospitalier de L'Universite de Montreal Hopital Notre-Dame, Montreal, Quebec
- Denmark (3):
  - Herlev og Gentofte Hospital, Herlev
  - Rigshospitalet, KÃ¸benhavn
  - Odense Universitetshospital, Odense C
- Finland (4):
  - Docrates Syopasairaala, Helsinki
  - Helsingin Yliopistollinen Keskussairaala, Helsinki
  - Oulu University Hospital, Oulu
  - Turku University Hospital, Turku
- France (18):
  - Centre Hospitalier Regional Universitaire - Hopital Morvan, Brest
  - Centre Hospitalier Intercommunal de CrÃ©teil, CrÃ©teil
  - Centre Hospitalier Universitaire de Grenoble - Hopital Nord Michallon, Grenoble
  - Centre Hospitalier Universitaire RÃ©gional de Lille - HÃ´pital Albert Calmette, Lille
  - Centre Hospitalier Universitaire de Limoges - Hopital Dupuytren, Limoges
  - Centre Leon Berard, Lyon
  - Centre Hospitalier Universitaire Nord, Marseille
  - Institut Curie, Paris
  - Hopital Cochin, Paris
  - Hopital Bichat Claude Bernard, Paris
  - HÃ´pital Tenon, Paris
  - Centre Hospitalier Universitaire de Bordeaux - Hopital Haut Leveque, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Hospitalier Universitaire de Rennes - Hopital Pontchaillou, Rennes
  - Centre Hospitalier de Nantes - HÃ´pital Nord LaÃ"nnec, Saint-Herblain
  - Centre Hospitalier Universitaire de Strasbourg - Nouvel Hopital Civil, Strasbourg
  - Centre Hospitalier Universitaire de Toulouse - Hopital Larrey, Toulouse
  - Gustave Roussy, Villejuif
- Germany (15):
  - Evangelische Lungenklinik, Berlin
  - Charite UniversitÃ¤tsmedizin Berlin, CharitÃ© Campus Virchow-Klinikum, Berlin
  - Universitaetsklinikum Carl Gustav Carus, Dresden
  - UniversitÃ¤tsklinikum Essen, Essen
  - Klinikum Esslingen GmbH, Esslingen am Neckar
  - UniversitÃ¤tsklinikum Frankfurt/Main, Frankfurt am Main
  - Asklepios - Fachkliniken MÃ¼nchen-Gauting, Gauting
  - LungenClinic Grosshansdorf GmbH, Großhansdorf
  - Studiengesellschaft HÃ¤mato Onkologie Hamburg Prof Laack und Partner, Hamburg
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Klinikverbund AllgÃ¤u, Immenstadt im Allgäu
  - Universitatsklinikum Koln, KÃ¶ln
  - Pneumologisch/onkologisch/internistisches Studienzentrum, Leipzig
  - Bethanien Krankenhaus, Moers
  - Pius-Hospital Oldenburg, Oldenburg
- Greece (12):
  - Agios Savvas Anticancer Hospital, Athens
  - Henry Dunant Hospital Center, Athens
  - Sotiria General Hospital, Athens
  - General Oncology Hospital of Kifissia Agioi Anargyroi, Athens
  - Metropolitan Hospital, Athens
  - University Hospital of Heraklion, Heraklion - Crete
  - University Hospital of Larissa, Larissa
  - University Hospital of Patras, Pátrai
  - Theagenion Cancer Hospital, Thessaloniki
  - Bioclinic of Thessaloniki, Thessaloniki
  - Euromedica General Clinic of Thessaloniki, Thessaloniki
  - Agios Loukas Clinic, Thessaloniki
- Hungary (9):
  - Semmelweis Egyetem, Budapest
  - Orszagos Koranyi Pulmonologiai Intezet, Budapest
  - Veszprem Megyei Tudogyogyintezet, Farkasgyepű
  - Bekes Megyei Kozponti Korhaz Pandy Kalman Tagkorhaz, Gyula
  - Somogy Megyei Kaposi Mor Oktato Korhaz, Kaposvár
  - Borsod-Abauj-Zemplen Megyei Kozponti Korhaz es Egyetemi Oktatokorhaz, Miskolc
  - Fejer Megyei Szent Gyorgy Egyetemi Oktato Korhaz, Székesfehérvár
  - Szent Borbala Korhaz, Tatabánya
  - Tudogyogyintezet Torokbalint, Törökbálint
- Italy (16):
  - Azienda Ospedaliera di Rilievo Nazionale San Giuseppe Moscati, Avellino
  - IRCCS Istituto Tumori Giovanni Paolo II, Bari
  - Azienda Ospedaliera Universitaria di Bologna Policlinico S Orsola Malpighi, Bologna
  - Azienda Ospedaliera Universitaria Policlinico Vittorio Emanuele Presidio Ospedaliero G Rodolico, Catania
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Azienda Ospedaliero Universitaria di Cagliari Policlinico Duilio Casula, Monserrato CA
  - Azienda Socio Sanitaria Territoriale di Monza Ospedale San Gerardo, Monza (MB)
  - Azienda Ospedaliera di Rilievo Nazionale Specialistica dei Colli Monaldi, Napoli
  - Azienda Ospedaliera Universitaria San Luigi Gonzaga, Orbassano (TO)
  - Istituto Oncologico Veneto IRCCS, Padua
  - Azienda UnitÃ Sanitaria Locale della Romagna Presidio ospedaliero di Ravenna, Ravenna
  - Azienda Ospedaliera Policlinico Umberto I, Roma
  - Policlinico Universitario Agostino Gemelli, Roma
- Japan (40):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Chiba Cancer Center, Chiba, Chiba
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - National Hospital Organization Kyushu Cancer Center, Fukuoka, Fukuoka
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Hospital of the University of Occupational and Environmental Health, Kitakyushu-shi, Fukuoka
  - Chugoku Central Hospital of Japan Mutual Aid Association of Public School Teachers, Fukuyama-shi, Hiroshima
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - National Hospital Organization Hokkaido Cancer Center, Sapporo, Hokkaido
  - Hyogo Cancer Center, Akashi-shi, Hyōgo
  - National Hospital Organization Himeji Medical Center, Himeji-shi, Hyōgo
  - Itami City Hospital, Itami-shi, Hyōgo
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - St Marianna University School of Medicine Hospital, Kawasaki-shi, Kanagawa
  - Kitasato University Hospital, Sagamihara-shi, Kanagawa
  - Kanagawa Prefectural Hospital Organization Kanagawa Cancer Center, Yokohama, Kanagawa
  - Kyoto University Hospital, Kyoto, Kyoto
  - Miyagi Cancer Center, Natori-shi, Miyagi
  - Sendai Kousei Hospital, Sendai, Miyagi
  - Niigata Cancer Center Hospital, Niigata, Niigata
  - Okayama University Hospital, Okayama, Okayama-ken
  - Osaka Habikino Medical Center, Habikino-shi, Osaka
  - Kansai Medical University Hospital, Hirakata-shi, Osaka
  - Osaka City General Hospital, Osaka, Osaka
  - Osaka International Cancer Institute, Osaka, Osaka
  - Kindai University Hospital, Osakasayama-shi, Osaka
  - National Hospital Organization Kinki-chuo Chest Medical Center, Sakai-shi, Osaka
  - Saga-ken Medical Centre Koseikan, Saga, Saga-ken
  - Saitama Cancer Center, Kitaadachi-gun, Saitama
  - Shiga University of Medical Science Hospital, Ōtsu, Shiga
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Cancer Institute Hospital of Japanese Foundation for Cancer Research, Koto-ku, Tokyo
  - Tottori University Hospital, Yonago-shi, Tottori
  - Wakayama Medical University Hospital, Wakayama, Wakayama
  - National Hospital Organization Iwakuni Clinical Center, Iwakuni-shi, Yamaguchi
  - National Hospital Organization Yamaguchi Ube Medical Center, Ube-shi, Yamaguchi
- Netherlands (5):
  - Nederlands Kanker Instituut Antoni van Leeuwenhoekziekenhuis, Amsterdam
  - Universitair Medisch Centrum Groningen, Groningen
  - Radboudumc, Nijmegen
  - Erasmus Medisch Centrum, Rotterdam
  - Universitair Medisch Centrum Utrecht, Utrecht
- Poland (5):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Instytut Genetyki i Immunologii GENIM Spzoo, Lublin
  - Szpital Kliniczny Przemienienia Panskiego Uniwersytetu Medycznego im K Marcinkowskiego w Poznaniu, Poznan
  - Centrum Onkologii Instytut im Marii Sklodowskiej-Curie, Warsaw
  - Dolnoslaskie Centrum Onkologii we Wroclawiu, Wroclaw
- Portugal (5):
  - Centro Hospitalar Universitario de Lisboa Norte EPE - Hospital Pulido Valente, Lisbon
  - Unidade Local de Saude de Matosinhos, EPE - Hospital Pedro Hispano, Matosinhos Municipality
  - Centro Hospitalar Universitario do Porto EPE - Hospital de Santo Antonio, Porto
  - Instituto Portugues de Oncologia do Porto Francisco Gentil, EPE, Porto
  - Centro Hospitalar Universitario de Sao Joao EPE - Hospital Sao Joao, Porto
- Russia (5):
  - Clinical hospital 2, Group of companies medsi, Moscow
  - LLC Tonus, Nizhny Novgorod
  - Omsk Regional Clinical Oncology Dispensary, Omsk
  - FSBI Scientific and Research Oncology Institute named after N N Petrov, Saint Petersburg
  - Saint Petersburg scientifical practical center of specialized kinds of medical care oncological, Saint Petersburg
- South Korea (11):
  - Chungbuk National University Hospital, Cheongju-si, Chungcheongbuk-do
  - National Cancer Center, Goyang-si Gyeonggi-do
  - Cha Bundang Medical Center, Cha University, Seongnam-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung medical center, Seoul
  - The Catholic University of Korea Seoul St Marys Hospital, Seoul
  - Ulsan University Hospital, Ulsan
- Spain (12):
  - Hospital Regional Universitario de Malaga, Málaga, AndalucÃ-a
  - Hospital Universitario Insular de Gran Canaria, Las Palmas de Gran Canaria, Canary Islands
  - Hospital Universitari Vall d Hebron, Barcelona, CataluÃ±a
  - Hospital Clinic i Provincial de Barcelona, Barcelona, CataluÃ±a
  - Hospital de la Santa Creu i Sant Pau, Barcelona, CataluÃ±a
  - Instituto Catalan de Oncologia Hospital Duran i Reynals, L'Hospitalet de Llobregat, CataluÃ±a
  - Complexo Hospitalario Universitario A CoruÃ±a Hospital Teresa Herrera, A CoruÃ±a, Galicia
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital Clinico Universitario de Valencia, Valencia, Valencia
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
- Sweden (6):
  - Gavle Sjukhus, Gävle
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Universitetssjukhuset i Linkoping, Linköping
  - Skanes Universitetssjukhus, Lund
  - Karolinska Universitetssjukhuset Solna, Stockholm
  - Norrlands Universitetssjukhus, Umeå
- Switzerland (6):
  - Universitaetsspital Basel, Basel
  - Inselspital Bern, Bern
  - Hopitaux Universitaires de Geneve, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital Winterthur, Winterthur
  - Universitaetsspital Zuerich, Zurich
- Taiwan (4):
  - China Medical University Hospital, Taichung
  - Veterans General Hospital - Taichung, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
- United Kingdom (8):
  - Addenbrookes Hospital, Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Western General Hospital, Edinburgh
  - Royal Marsden Hospital, London
  - Sarah Cannon Research Institute UK, London
  - Christie Hospital, Manchester
  - Nottingham City Hospital, Nottingham
  - Churchill Hospital, Oxford
  - Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] Waterhouse DM, Rothschild S, Dooms C, Mennecier B, Bozorgmehr F, Majem M, van den Heuvel MH, Linardou H, Chul Cho B, Roberts-Thomson R, Tanaka K, Blais N, Schvartsman G, Holmskov Hansen K, Chmielewska I, Forster MD, Giannopoulou C, Stollenwerk B, Obiozor CC, Wang Y, Novello S. Patient-reported outcomes in CodeBreaK 200: Sotorasib versus docetaxel for previously treated advanced NSCLC with KRAS G12C mutation. Lung Cancer. 2024 Oct;196:107921. doi: 10.1016/j.lungcan.2024.107921. Epub 2024 Aug 6. PMID 39303400
- [Background] Skoulidis F, Li BT, Hochmair M, Govindan R, Vincent M, van der Wekken AJ, Reguart Aransay N, O'Byrne KJ, Girard N, Griesinger F, Nishio M, Hafliger S, Lindsay C, Reinmuth N, Paulus A, Papakotoulas P, Kim SW, Ferreira CG, Pasello G, Duruisseaux M, Gennatas S, Dimou A, Mehta B, Kormany W, Nduka C, Sylvester BE, Ardito-Abraham C, Wang Y, de Langen AJ. Pooled safety analysis and management of sotorasib-related adverse events in KRAS G12C-mutated advanced non-small cell lung cancer. Oncologist. 2025 Jan 17;30(1):oyae356. doi: 10.1093/oncolo/oyae356. PMID 39846981
- [Background] Skoulidis F, Li BT, de Langen AJ, Hong DS, Lena H, Wolf J, Dy GK, Curioni Fontecedro A, Tomasini P, Velcheti V, van der Wekken AJ, Dooms C, Paz-Ares Rodriguez L, Mountzios G, Sacher A, Nadal E, Couraud S, Kim SW, O'Byrne K, Rocco D, Toyozawa R, Chmielewska I, Lindsay CR, Hindoyan A, Mukundan L, Wilmanski T, Anderson A, Ardito-Abraham C, Pati A, Reddy A, Mehta B, Schuler M. Molecular determinants of sotorasib clinical efficacy in KRASG12C-mutated non-small-cell lung cancer. Nat Med. 2025 Aug;31(8):2755-2767. doi: 10.1038/s41591-025-03732-5. Epub 2025 May 28. PMID 40437272
- [Background] de Langen AJ, Johnson ML, Mazieres J, Dingemans AC, Mountzios G, Pless M, Wolf J, Schuler M, Lena H, Skoulidis F, Yoneshima Y, Kim SW, Linardou H, Novello S, van der Wekken AJ, Chen Y, Peters S, Felip E, Solomon BJ, Ramalingam SS, Dooms C, Lindsay CR, Ferreira CG, Blais N, Obiozor CC, Wang Y, Mehta B, Varrieur T, Ngarmchamnanrith G, Stollenwerk B, Waterhouse D, Paz-Ares L; CodeBreaK 200 Investigators. Sotorasib versus docetaxel for previously treated KRAS G12C-mutated non-small-cell lung cancer: a plain language summary. Future Oncol. 2025 Apr;21(9):1033-1044. doi: 10.1080/14796694.2025.2474789. Epub 2025 Mar 24. Erratum In: Future Oncol. PMID 40129223
- [Background] Dingemans AC, Syrigos K, Livi L, Paulus A, Kim SW, Chen Y, Felip E, Griesinger F, Ohashi K, Zalcman G, Hughes BGM, Sorensen JB, Blais N, Ferreira CGM, Lindsay CR, Dziadziuszko R, Ward PJ, Obiozor CC, Wang Y, Peters S. Intracranial activity of sotorasib vs docetaxel in pretreated KRAS G12C-mutated advanced non-small cell lung cancer from a global, phase 3, randomized controlled trial. Lung Cancer. 2025 Sep;207:108683. doi: 10.1016/j.lungcan.2025.108683. Epub 2025 Jul 29. PMID 40774040
- [Derived] de Langen AJ, Johnson ML, Mazieres J, Dingemans AC, Mountzios G, Pless M, Wolf J, Schuler M, Lena H, Skoulidis F, Yoneshima Y, Kim SW, Linardou H, Novello S, van der Wekken AJ, Chen Y, Peters S, Felip E, Solomon BJ, Ramalingam SS, Dooms C, Lindsay CR, Ferreira CG, Blais N, Obiozor CC, Wang Y, Mehta B, Varrieur T, Ngarmchamnanrith G, Stollenwerk B, Waterhouse D, Paz-Ares L; CodeBreaK 200 Investigators. Sotorasib versus docetaxel for previously treated non-small-cell lung cancer with KRASG12C mutation: a randomised, open-label, phase 3 trial. Lancet. 2023 Mar 4;401(10378):733-746. doi: 10.1016/S0140-6736(23)00221-0. Epub 2023 Feb 7. PMID 36764316
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 345 participants were enrolled at 148 centers in Europe, North America, Asia, Australia, and South America. The analyses presented in this results summary are based on the primary completion data. The primary completion data cut-off was 02 August 2022. The study is ongoing.
Pre-assignment Details: Screening assessments were conducted within 28 days before Cycle 1 Day 1 (C1D1; where a cycle is 21 days). Participants were then randomized 1:1 to receive either AMG 510 or docetaxel, stratified by number of prior lines of therapy in advanced disease (1 vs 2 vs > 2), race (Asian vs non-Asian), and history of central nervous system (CNS) involvement (present or absent).
Groups:
- AMG 510: Participants with previously treated locally advanced and unresectable or metastatic non small cell lung cancer (NSCLC) with centrally confirmed Kirsten rat sarcoma viral oncogene homolog (KRAS) p.G12C mutation received 960 mg of AMG 510 orally via tablets once a day (QD) in each 21 day cycle.
- Docetaxel: Participants with previously treated locally advanced and unresectable or metastatic NSCLC with centrally confirmed KRAS p.G12C mutation received 75 mg/m^2 of docetaxel via intravenous (IV) infusion once every 3 weeks (Q3W) in each 21 day cycle. Participants who were determined to have radiological progression according to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) by the investigator and progressive disease confirmed by independent central imaging review, could have switched to receive AMG 510. Alternatively, if an early efficacy of the study is noted by the data monitoring committee, crossover would be considered for all participants who randomized into the docetaxel arm (so that they are able to immediately receive AMG 510).
Period: Overall Study
Arm/Group | AMG 510 | Docetaxel
Started | 171 | 174
Switched From Docetaxel to AMG 510 | 0 | 46
Completed (Number of participants who have completed the study as of the primary analysis completion date (02 August 2022).) | 0 | 3
Not Completed | 171 | 171
Not completed — Death | 104 | 85
Not completed — Lost to Follow-up | 5 | 2
Not completed — Withdrawal by Subject | 12 | 39
Not completed — Ongoing in study | 50 | 45

BASELINE CHARACTERISTICS:
Population: As pre-specified in the statistical analysis plan, data are presented for all randomized participants according to original treatment assignment, regardless of whether participants switched from receiving docetaxel to receiving AMG 510.
Groups:
- AMG 510: Participants with previously treated locally advanced and unresectable or metastatic NSCLC with centrally confirmed KRAS p.G12C mutation received 960 mg of AMG 510 orally via tablets QD in each 21 day cycle.
- Total: Total of all reporting groups
Arm/Group | AMG 510 | Docetaxel | Total
Number analyzed (Participants) | 171 | 174 | 345
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (9.9) | 63.6 (9.1) | 63.5 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 79 | 141
  Male | 109 | 95 | 204
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 9 | 14
  Not Hispanic or Latino | 165 | 163 | 328
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 21 | 22 | 43
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 142 | 144 | 286
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 5 | 8 | 13

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from randomization (baseline) until disease progression or death from any cause, whichever occurred first for all participants. Progression was based on blinded independent central review (BICR) of disease response per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).
  As pre-specified in the statistical analysis plan, for participants who crossed over from docetaxel to AMG 510, the participant's response post first progression or post crossover was not used for the primary analyses. Data are presented per original treatment randomized.
Time Frame: Baseline up to primary analysis data cut-off date (02 August 2022); max time on study as of primary analysis data cut off was 24.3 months
Population: Measured in the Full Analysis Set (FAS), which included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AMG 510 | Docetaxel
Number analyzed (Participants) | 171 | 174
months | 5.62 [4.27 to 7.75] | 4.47 [3.02 to 5.68]
Statistical Analysis 1: Comparison: AMG 510 vs Docetaxel; Test type: Equivalence — A hazard ratio <1.0 indicates a lower average event rate and a longer PFS for AMG 510 relative to docetaxel. P-value was calculated using a stratified log-rank test; p = 0.002, Log Rank; Hazard Ratio (HR) = 0.663, 95% CI 2-sided [0.509 to 0.864]

ADVERSE EVENTS:
Time Frame: Adverse events:for 'Docetaxel' and 'AMG 510', from first dose(FD) to 30 days post last dose, or before FD of AMG 510 if participants cross over, or end of study (EOS) or data cut-off (DCO) which occurred earliest; median[min,max] duration 4.06[0.2,23.7] mons. For 'Docetaxel, then Switched to AMG 510', from FD to EOS/DCO which occurred earliest; median[min,max] duration 7.97[0.8,15.2] mons. Mortality:from randomization until death or DCO; median[min,max] time on study 14.78[0.2,24.3] mons.
Description: Serious and other adverse events are reported for all participants who received at least one dose of study drug. All-cause mortality is reported for all randomized participants. As pre-specified in the statistical analysis plan, data are reported per treatment received, including participants who were randomized to docetaxel and switched to AMG 510.
Groups:
- Docetaxel, Then Switched to AMG 510: Participants who were randomized to originally receive docetaxel, who were determined to have radiological progression according to RECIST v1.1 by the investigator and progressive disease confirmed by independent central imaging review, and switched to receive AMG 510. Alternatively, participants could switch from docetaxel to receive AMG 510 if an early efficacy of the study is noted by the data monitoring committee.
Arm/Group | Docetaxel | AMG 510 | Docetaxel, Then Switched to AMG 510
All-Cause Mortality (participants affected / at risk) | 78/174 | 109/171 | 17/46
Serious Adverse Events (participants affected / at risk) | 67/151 | 91/169 | 26/46
Other Adverse Events (participants affected / at risk) | 129/151 | 151/169 | 35/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel (N=151) | AMG 510 (N=169) | Docetaxel, Then Switched to AMG 510 (N=46)
Anaemia (Blood and lymphatic system disorders) | 5 | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 7 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Myocarditis (Cardiac disorders) | 0 | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Adrenal cortex necrosis (Endocrine disorders) | 1 | 0 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 3 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 5 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 2
Obstruction gastric (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 2 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0
Chest pain (General disorders) | 0 | 3 | 0
Fatigue (General disorders) | 2 | 0 | 0
General physical health deterioration (General disorders) | 1 | 1 | 0
Malaise (General disorders) | 2 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 1 | 0
Oedema peripheral (General disorders) | 1 | 1 | 0
Pain (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 2 | 3 | 0
Biliary obstruction (Hepatobiliary disorders) | 0 | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 2 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 1 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 2 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0
Appendicitis perforated (Infections and infestations) | 0 | 1 | 0
Atypical pneumonia (Infections and infestations) | 1 | 0 | 0
Bacterial diarrhoea (Infections and infestations) | 1 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 1 | 2 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0
Infection (Infections and infestations) | 1 | 2 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0
Peritonitis (Infections and infestations) | 0 | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 2 | 0 | 0
Pneumonia (Infections and infestations) | 10 | 1 | 2
Pneumonia aspiration (Infections and infestations) | 2 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 1 | 0
Pneumonia legionella (Infections and infestations) | 1 | 0 | 0
Pneumonia pneumococcal (Infections and infestations) | 1 | 0 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 3 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Urinary tract infection bacterial (Infections and infestations) | 0 | 1 | 0
Wound infection staphylococcal (Infections and infestations) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound secretion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 0
General physical condition abnormal (Investigations) | 0 | 1 | 0
Liver function test increased (Investigations) | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 1
Food intolerance (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 18 | 9
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1
Non-small cell lung cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Tumour hyperprogression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Altered state of consciousness (Nervous system disorders) | 1 | 0 | 0
Aphasia (Nervous system disorders) | 1 | 0 | 0
Cerebellar syndrome (Nervous system disorders) | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0
Paraplegia (Nervous system disorders) | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0
Seizure (Nervous system disorders) | 1 | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 1
Thrombotic stroke (Nervous system disorders) | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Renal injury (Renal and urinary disorders) | 0 | 0 | 1
Oedema genital (Reproductive system and breast disorders) | 0 | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Paraneoplastic pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0
Mucocutaneous rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
Intermittent claudication (Vascular disorders) | 1 | 0 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel (N=151) | AMG 510 (N=169) | Docetaxel, Then Switched to AMG 510 (N=46)
Anaemia (Blood and lymphatic system disorders) | 30 | 28 | 5
Neutropenia (Blood and lymphatic system disorders) | 14 | 3 | 2
Abdominal pain (Gastrointestinal disorders) | 9 | 20 | 3
Abdominal pain upper (Gastrointestinal disorders) | 5 | 11 | 3
Constipation (Gastrointestinal disorders) | 29 | 22 | 3
Diarrhoea (Gastrointestinal disorders) | 37 | 70 | 14
Nausea (Gastrointestinal disorders) | 36 | 43 | 6
Stomatitis (Gastrointestinal disorders) | 19 | 3 | 0
Vomiting (Gastrointestinal disorders) | 15 | 22 | 2
Asthenia (General disorders) | 21 | 16 | 4
Chest pain (General disorders) | 2 | 12 | 2
Fatigue (General disorders) | 43 | 27 | 6
Malaise (General disorders) | 9 | 4 | 0
Mucosal inflammation (General disorders) | 11 | 1 | 0
Oedema (General disorders) | 8 | 3 | 0
Oedema peripheral (General disorders) | 19 | 4 | 2
Pain (General disorders) | 9 | 6 | 2
Pyrexia (General disorders) | 18 | 8 | 1
COVID-19 (Infections and infestations) | 5 | 2 | 5
Alanine aminotransferase increased (Investigations) | 1 | 17 | 4
Aspartate aminotransferase increased (Investigations) | 1 | 17 | 3
Blood alkaline phosphatase increased (Investigations) | 3 | 13 | 3
Weight decreased (Investigations) | 7 | 9 | 2
Decreased appetite (Metabolism and nutrition disorders) | 29 | 39 | 5
Hypoalbuminaemia (Metabolism and nutrition disorders) | 8 | 4 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 12 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 8 | 5 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 | 26 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 23 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 9 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 8 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 15 | 8 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 11 | 2
Dizziness (Nervous system disorders) | 7 | 10 | 3
Dysgeusia (Nervous system disorders) | 14 | 4 | 0
Headache (Nervous system disorders) | 13 | 12 | 2
Neuropathy peripheral (Nervous system disorders) | 16 | 1 | 0
Insomnia (Psychiatric disorders) | 8 | 9 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 25 | 22 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 25 | 30 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 35 | 3 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 15 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2022-01-06): https://cdn.clinicaltrials.gov/large-docs/80/NCT04303780/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-21): https://cdn.clinicaltrials.gov/large-docs/80/NCT04303780/SAP_001.pdf